CLINICAL TRIAL: NCT00453921
Title: Methylphenidate (Ritalin) and Memory/Attention in Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laura Flashman, Professor of Psychiatry, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17363; 5R01HD047242 (NIH)
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Brain Injury
Keywords: TBI; Memory; Methylphenidate; Ritalin; Memory and Attention Training
MeSH Terms: conditions — Brain Injuries | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Placebo Capsule and Placebo Memory and Attention Training (Placebo as both conditions)
  Interventions: Other: Placebo as both treatments
- 2 (Active Comparator): Methylphenidate capsules and Memory and Attention Training (Active Med/Active therapy)
  Interventions: Drug: Methylphenidate; Behavioral: Memory and Attention Training
- 3 (Active Comparator): Methylphenidate capsules and Placebo Memory and Attention Training (Active Med/Placebo therapy)
  Interventions: Drug: Methylphenidate
- 4 (Active Comparator): Placebo capsules and Memory and Attention Training (Placebo Med/Active therapy)
  Interventions: Behavioral: Memory and Attention Training

INTERVENTIONS:
Drug: Methylphenidate — Dosage dependent on weight
  Arms: 2; 3
Behavioral: Memory and Attention Training — Weekly Memory and Attention Training with at home practice.
  Arms: 2; 4
Other: Placebo as both treatments — Placebo capsules and Placebo Memory and Attention Training
  Arms: 1

SUMMARY:
Traumatic brain injury (TBI) is a significant public health problem, with 1.5-2.0 million Americans injured each year. Cognitive deficits, particularly in the domains of memory and attention are frequently the source of lingering disability after TBI and a source of enormous distress to the injured individuals and their family/caregivers. To date, interventions to ameliorate chronic cognitive deficits have been directed at either pharmacological interventions or cognitive rehabilitation. We propose to (1) To compare the efficacy of three interventions: memory and attention training (MAAT), methylphenidate, and memory/attention training in combination with methylphenidate and (2) use functional MRI (fMRI) to characterize changes in activation of the neural circuitry of memory and attention due to MAAT alone, methylphenidate alone, and MAAT in combination with methylphenidate. This is a two by two design with medication (methylphenidate/placebo) and cognitive therapy (Memory and Attention Training (MAAT) or an Attention control intervention) as possible interventions. Using a randomized, placebo-controlled, double-blind design, 200 individuals with persistent cognitive deficits 6-12 months after MTBI will be randomized to receive a six week trial of either (1) MAAT and placebo, (2) MAAT and methylphenidate (0.3 mg/kg BID), (3) attention control intervention and methylphenidate (0.3 mg/kg BID), or (4) attention control intervention and placebo. Symptom distress, attention and memory performance, and activation patterns of the neural circuitry of attention and memory while undergoing fMRI will be characterized at baseline, and after the four treatment conditions. This study will provide important information on three interventions for the most disabling sequelae of an enormous public health problem. Further, it will help to clarify underlying neural mechanisms and suggest additional treatment possibilities.

DETAILED DESCRIPTION:
Summary and Gaps to be Addressed by the Proposed Study

What is known: There are two interventions of promising efficacy in ameliorating deficits in attention and memory after mild traumatic brain injury (MTBI): (i) memory and attention training/rehabilitation, and (ii) catecholaminergic augmentation (particularly with methylphenidate - which augments both dopaminergic and adrenergic systems). fMRI and other functional imaging strategies are providing valuable insights into the underlying neural mechanisms of the cognitive enhancing effects of methylphenidate in some neuropsychiatric populations (individuals with ADHD), and the effects of cognitive rehabilitation efforts in some domains (e.g. speech and language in individuals after stroke).

What is not known: To date there are no studies that apply a psychopharmacological strategy of augmenting neurotransmitter systems known to modulate memory/attention (dopaminergic and adrenergic systems) in combination with a cognitive rehabilitation intervention known to improve memory/attention (memory/attention training) in individuals with MTBI. We are aware of no published studies that use fMRI to assess the neural mechanisms of memory/attention improvement from the use of catecholaminergic agents or memory/attention training in individuals with MTBI. It is important to determine the efficacy of combined memory/attention training and methylphenidate. It is equally important to begin to understand the neural mechanisms underlying effective treatment as it may help to inform the development of the next generation of interventions and perhaps lead to individually tailored treatment interventions. This proposal will start to address these gaps in our knowledge.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Individuals aged 18-65 who sustained a mild to severe TBI 4 months prior to study entry.
2. TBI: Subjects must sustain a traumatic blow to the head, resulting in either alteration of level of consciousness (manifested by being dazed and confused or having amnesia for the event) or loss of consciousness (LOC). Duration of LOC will be estimated by using all available information including patient and witness reports, emergency personnel records and Dartmouth Hitchcock Medical Center (DHMC) medical records. Post traumatic amnesia (PTA) will be estimated by careful questioning of patients to determine the time of return of continuous memory. This will be informed by review of medical records. We plan to include individuals with intracranial or skull injuries stemming from the TBI, providing they meet the inclusion criteria. Such lesions will be catalogued, and included as a factor in the data analysis.
3. Cognitive Deficits: Subjects will have either subjective and objective evidence of persistent cognitive deficits. Subjects must report persistent memory or attention deficits as a result of their injury, which are of sufficient severity to interfere with social and/or occupational functioning. Subjects must either score more than 2 standard deviations below the age adjusted norm or estimates of baseline premorbid function on one or more tests of attention and/or memory administered as part of the baseline screening cognitive battery (see below), or score greater than 1.0 standard deviations below either age adjusted norms or estimates of premorbid function on 2 or more of the screening tests.

Exclusion Criteria:

The following factors will exclude otherwise eligible subjects from participation:

1. a history of other neurologic disorders (such as epilepsy, cerebrovascular disease, mental retardation, neurodegenerative disorders)
2. significant systemic medical illness such as clinically significant liver disease, renal disease, atherosclerotic coronary vascular disease, or hypertension requiring medication management
3. current Diagnostic and Statistical Manual (DSM-IV) Axis I diagnosis of psychiatric illness other than substance abuse. We have given careful consideration to the inclusion of the latter group given our use of a stimulant with potential abuse properties. Because of the potential for cross-over abuse with cocaine, amphetamines, and other stimulants, individuals with such histories will be excluded from this study. Individuals with history of otherwise uncomplicated ethanol or other non-stimulant drug abuse currently in stable remission will be eligible. The Structured Clinical Interview for DSM-IV (MINI) will be used to screen for psychiatric illness
4. women currently pregnant or lactating. Female participants will be asked to take a pregnancy test to confirm they are not currently pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W McAllister, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center, Dartmouth Medical School
Locations (3):
- United States (3):
  - University of Colorado at Denver, Denver, Colorado
  - Indiana University, Indianapolis, Indiana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Background] McAllister TW, Flashman LA, McDonald BC, Saykin AJ. Mechanisms of working memory dysfunction after mild and moderate TBI: evidence from functional MRI and neurogenetics. J Neurotrauma. 2006 Oct;23(10):1450-67. doi: 10.1089/neu.2006.23.1450. PMID 17020482
- [Background] Neurobehavioral Guidelines Working Group; Warden DL, Gordon B, McAllister TW, Silver JM, Barth JT, Bruns J, Drake A, Gentry T, Jagoda A, Katz DI, Kraus J, Labbate LA, Ryan LM, Sparling MB, Walters B, Whyte J, Zapata A, Zitnay G. Guidelines for the pharmacologic treatment of neurobehavioral sequelae of traumatic brain injury. J Neurotrauma. 2006 Oct;23(10):1468-501. doi: 10.1089/neu.2006.23.1468. PMID 17020483
- [Background] McAllister TW, Rhodes CH, Flashman LA, McDonald BC, Belloni D, Saykin AJ. Effect of the dopamine D2 receptor T allele on response latency after mild traumatic brain injury. Am J Psychiatry. 2005 Sep;162(9):1749-51. doi: 10.1176/appi.ajp.162.9.1749. PMID 16135640
- [Background] McAllister TW, Flashman LA, Sparling MB, Saykin AJ. Working memory deficits after traumatic brain injury: catecholaminergic mechanisms and prospects for treatment -- a review. Brain Inj. 2004 Apr;18(4):331-50. doi: 10.1080/02699050310001617370. PMID 14742148
- [Background] McAllister TW, Ferrell RB. Evaluation and treatment of psychosis after traumatic brain injury. NeuroRehabilitation. 2002;17(4):357-68. PMID 12547983
- [Background] Flashman LA, McAllister TW. Lack of awareness and its impact in traumatic brain injury. NeuroRehabilitation. 2002;17(4):285-96. PMID 12547977
- [Background] McAllister TW, Arciniegas D. Evaluation and treatment of postconcussive symptoms. NeuroRehabilitation. 2002;17(4):265-83. PMID 12547976
- [Background] McAllister TW. Evaluation and treatment of neurobehavioral complications of traumatic brain injury--have we made any progress? NeuroRehabilitation. 2002;17(4):263-4. No abstract available. PMID 12547975
- [Background] McAllister TW, Sparling MB, Flashman LA, Saykin AJ. Neuroimaging findings in mild traumatic brain injury. J Clin Exp Neuropsychol. 2001 Dec;23(6):775-91. doi: 10.1076/jcen.23.6.775.1026. PMID 11910544
- [Background] McAllister TW, Sparling MB, Flashman LA, Guerin SJ, Mamourian AC, Saykin AJ. Differential working memory load effects after mild traumatic brain injury. Neuroimage. 2001 Nov;14(5):1004-12. doi: 10.1006/nimg.2001.0899. PMID 11697932
- [Background] McAllister TW, Saykin AJ, Flashman LA, Sparling MB, Johnson SC, Guerin SJ, Mamourian AC, Weaver JB, Yanofsky N. Brain activation during working memory 1 month after mild traumatic brain injury: a functional MRI study. Neurology. 1999 Oct 12;53(6):1300-8. doi: 10.1212/wnl.53.6.1300. PMID 10522888
- [Background] McAllister TW. Traumatic Brain Injury and Psychosis: What Is the Connection? Semin Clin Neuropsychiatry. 1998 Jul;3(3):211-223. PMID 10085209
- [Background] Flashman LA, Amador X, McAllister TW. Lack of Awareness of Deficits in Traumatic Brain Injury. Semin Clin Neuropsychiatry. 1998 Jul;3(3):201-210. PMID 10085208
- [Background] McAllister TW, Green RL. Traumatic Brain Injury: A Model of Acquired Psychiatric Illness? Semin Clin Neuropsychiatry. 1998 Jul;3(3):158-159. No abstract available. PMID 10085203
- [Background] McAllister TW. Evaluation of brain injury related behavioral disturbances in community mental health centers. Community Ment Health J. 1997 Aug;33(4):341-58; discussion 359-64. doi: 10.1023/a:1025055426260. PMID 9250431
- [Background] Silver JM, McAllister TW. Forensic issues in the neuropsychiatric evaluation of the patient with mild traumatic brain injury. J Neuropsychiatry Clin Neurosci. 1997 Winter;9(1):102-13. doi: 10.1176/jnp.9.1.102. No abstract available. PMID 9017537
- [Background] McAllister TW. Neuropsychiatric sequelae of head injuries. Psychiatr Clin North Am. 1992 Jun;15(2):395-413. PMID 1603732
- See also: Brain Injury Association of New Hampshire — http://www.bianh.org
- See also: Brain Injury Association of Vermont — http://www.biavt.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Both Conditions: Placebo Capsule and Placebo Memory and Attention Training (Placebo as both conditions)
  Placebo as both treatments: Placebo capsules and Placebo Memory and Attention Training
- Active Drug/Active Therapy: Methylphenidate capsules and Memory and Attention Training (Active Med/Active therapy)
  Methylphenidate: Dosage dependent on weight
  Memory and Attention Training: Weekly Memory and Attention Training with at home practice.
- Active Drug/Placebo Therapy: Methylphenidate capsules and Placebo Memory and Attention Training (Active Med/Placebo therapy)
  Methylphenidate: Dosage dependent on weight
- Placebo Drug/Active Therapy: Placebo capsules and Memory and Attention Training (Placebo Med/Active therapy)
  Memory and Attention Training: Weekly Memory and Attention Training with at home practice.
Period: Overall Study
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy
Started | 19 | 18 | 20 | 19
Completed | 18 | 17 | 18 | 18
Not Completed | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Individuals age 18-65 with a traumatic brain injury of at least mild severity at least 4 months prior to study entry, with self-report of cognitive deficits as a result of the injury of sufficient severity to interfere with social and/or occupational functioning.
Groups:
- Placebo Both Conditions: Placebo as both treatments: Placebo capsules and Placebo Memory and Attention Training
- Active Drug/Active Therapy: Methylphenidate: Dosage dependent on weight
  Memory and Attention Training: Weekly Memory and Attention Training with at home practice.
- Active Drug/Placebo Therapy: Methylphenidate: Dosage dependent on weight
- Placebo Drug/Active Therapy: Memory and Attention Training: Weekly Memory and Attention Training with at home practice.
- Total: Total of all reporting groups
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy | Total
Number analyzed (Participants) | 19 | 18 | 20 | 19 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant withdrew from study
  years
    number analyzed (Participants) | 19 | 18 | 20 | 18 | 75
    (all) | 37.3 (14.2) | 43.1 (12.3) | 43.0 (15.0) | 37.2 (12.0) | 40.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant withdrew from study
  Participants
    number analyzed (Participants) | 19 | 18 | 20 | 18 | 75
    Female | 6 | 10 | 6 | 4 | 26
    Male | 13 | 8 | 14 | 14 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant discontinued participation
  Participants
    number analyzed (Participants) | 19 | 18 | 20 | 18 | 75
    Hispanic or Latino | 0 | 1 | 0 | 1 | 2
    Not Hispanic or Latino | 19 | 17 | 20 | 17 | 73
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant discontinued participation
  Participants
    number analyzed (Participants) | 19 | 18 | 20 | 18 | 75
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 1 | 0 | 2
    White | 19 | 17 | 19 | 17 | 72
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: One participant discontinued
  Participants
    United States: number analyzed (Participants) | 19 | 18 | 20 | 18 | 75
    United States | 19 | 18 | 20 | 18 | 75

OUTCOME MEASURES:

1. Primary Outcome: Neuropsychological Assessment, CVLT-II
Description: Memory measure: California Verbal Learning Test, 2nd edition (CVLT), Total, trials 1-5 (range: 0-80). Higher scores are better outcome.
Time Frame: post-intervention (at least 7 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy
Number analyzed (Participants) | 18 | 17 | 19 | 17
units on a scale | 51.3 (1.9) | 51.8 (2.1) | 51.9 (1.9) | 57.2 (2.0)
Statistical Analysis 1: Comparison: Placebo Both Conditions vs Active Drug/Active Therapy vs Active Drug/Placebo Therapy vs Placebo Drug/Active Therapy; Test type: Other; p < 0.04, Kruskal-Wallis — For active therapy/placebo relative to both placebo

2. Primary Outcome: Neuropsychological Assessment - CPT, Distractibility Condition (Reaction Time)
Description: Continuous Performance Test, Distractibility Condition (Reaction Time in msecs) (range: 0-800). Higher score is worse performance.
Time Frame: post-intervention (at least 7 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy
Number analyzed (Participants) | 18 | 17 | 19 | 18
units on a scale | 426.4 (15.3) | 394.7 (17.3) | 416.6 (15.9) | 413.0 (17.3)

3. Primary Outcome: Functional MRI Task Performance and Brain Activation (Change From Baseline to Post-treatment)
Description: Change in performance (percent correct,adjusted for guessing) from pre-(baseline) to post-treatment (approximately 7 weeks) for in-scanner n-back working memory task (Range: 0-100). Higher scores means better performance.
Time Frame: pre- to post-6 week treatment intervention (at least 7 weeks)
Measure: Mean (Standard Deviation); unit: percentage of correct targets (adjusted)
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy
Number analyzed (Participants) | 12 | 10 | 10 | 10
percentage of correct targets (adjusted) | -4.46 (30.8) | 4.69 (26.8) | 4.86 (29.5) | -0.36 (23.4)
Statistical Analysis 1: Comparison: Placebo Both Conditions vs Active Drug/Active Therapy vs Active Drug/Placebo Therapy vs Placebo Drug/Active Therapy; Test type: Equivalence — Looking for statistical difference, p < .01, between groups looking at change scores; p < 0.05, ANOVA

4. Primary Outcome: Change in Anterior Cingulate Gyrus Activation During Working Memory Processing (3-back > 0-back Condition) From Baseline to Post-intervention
Description: Change from pre- to post-treatment in brain activation in the anterior cingulate region of interest in arbitrary units provided by the SPM (statistical parametric mapping) program (range: unknown). Higher scores indicate greater increase in activation from pre- to post-treatment.
Time Frame: pre- to post-intervention (at least 7 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy
Number analyzed (Participants) | 12 | 10 | 10 | 10
units on a scale | -0.31 (.36) | 0.09 (.36) | 0.20 (.42) | 0.05 (.27)
Statistical Analysis 1: Comparison: Placebo Both Conditions vs Active Drug/Active Therapy vs Active Drug/Placebo Therapy vs Placebo Drug/Active Therapy; Test type: Equivalence — group differences; p < 0.05, ANCOVA

5. Primary Outcome: Change in Left Middle/Inferior Frontal Activation During Working Memory Processing (3-back > 0-back Condition) From Baseline to Post-intervention
Description: Change from pre- to post-treatment in brain activation in the left middle/inferior frontal region of interest in arbitrary units provided by the SPM (statistical parametric mapping) program (range: unknown). Higher scores indicate greater increase in activation from pre- to post-treatment.
Time Frame: pre- to post-treatment (at least 7 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy
Number analyzed (Participants) | 12 | 10 | 10 | 10
units on a scale | -0.16 (.20) | 0.04 (.15) | 0.07 (.24) | .10 (.21)

6. Primary Outcome: Change in Right Inferior Frontal Activation During Working Memory Processing (3-back > 0-back Condition) From Baseline to Post-intervention
Description: Change from pre- to post-treatment in brain activation in the right inferior frontal region of interest in arbitrary units provided by the SPM (statistical parametric mapping) program (range: unknown). Higher scores indicate greater increase in activation from pre- to post-treatment.
Time Frame: pre- to post-treatment (at least 7 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy
Number analyzed (Participants) | 12 | 10 | 10 | 10
units on a scale | -0.18 (.28) | 0.05 (.28) | .15 (.29) | .14 (.22)

7. Secondary Outcome: Self Report Questionnaire - MASQ
Description: The Multiple Abilities Questionnaire (self rating) is a questionnaire in which participants can identify deficits/complaints in the areas of language, visual perception, verbal memory, visual memory and attention and concentration. A total score is calculated; range is 30-130. Higher scores indicate greater level of complaints (worse outcome). For the purposes of this study, a score one standard deviation above the mean (102.7) indicated significant reported cognitive complaints.
Time Frame: post-intervention (at least 7 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Both Conditions | Active Drug/Active Therapy | Active Drug/Placebo Therapy | Placebo Drug/Active Therapy
Number analyzed (Participants) | 19 | 18 | 20 | 18
units on a scale | 116.4 (4.5) | 120.5 (4.8) | 114.1 (4.5) | 118.1 (4.8)
Statistical Analysis 1: Comparison: Placebo Both Conditions vs Active Drug/Active Therapy vs Active Drug/Placebo Therapy vs Placebo Drug/Active Therapy; Test type: Other; p < 0.01, ANCOVA
Statistical Analysis 2: Comparison: Placebo Both Conditions vs Active Drug/Active Therapy vs Active Drug/Placebo Therapy vs Placebo Drug/Active Therapy; Test type: Superiority; p < 0.05, ANCOVA — a priopr

ADVERSE EVENTS:
Time Frame: 6 years
Description: Physical Symptom Checklist was completed at each visit and phone call.
Groups:
- Active Med/Active Therapy: Methylphenidate capsules and Memory and Attention Training (Active Med/Active therapy)
  Methylphenidate: Dosage dependent on weight
  Memory and Attention Training: Weekly Memory and Attention Training with at home practice.
- Active Med/Placebo Therapy: Methylphenidate capsules and Placebo Memory and Attention Training (Active Med/Placebo therapy)
  Methylphenidate: Dosage dependent on weight
- Placebo Med/Active Therapy: Placebo capsules and Memory and Attention Training (Placebo Med/Active therapy)
  Memory and Attention Training: Weekly Memory and Attention Training with at home practice.
Arm/Group | Placebo Both Conditions | Active Med/Active Therapy | Active Med/Placebo Therapy | Placebo Med/Active Therapy
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 8/19 | 12/18 | 11/20 | 9/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Both Conditions (N=19) | Active Med/Active Therapy (N=18) | Active Med/Placebo Therapy (N=20) | Placebo Med/Active Therapy (N=18)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 7 (18) | 6 (14) | 2 (5)
headache (Nervous system disorders) | 6 (9) | 11 (20) | 7 (16) | 8 (12)
Insomnia (Nervous system disorders) | 5 (12) | 7 (14) | 4 (6) | 3 (6)
Nervousness (Psychiatric disorders) | 2 (4) | 7 (20) | 6 (15) | 2 (4)
loss of appetite (Gastrointestinal disorders) | 1 (2) | 8 (30) | 5 (18) | 3 (6)
palpitations (Cardiac disorders) | 1 (1) | 4 (5) | 5 (5) | 1 (1)
dry mouth (General disorders) | 0 (0) | 2 (5) | 3 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (6) | 5 (9) | 5 (11) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 4 (6) | 4 (5) | 3 (4)
Depressed mood (Psychiatric disorders) | 3 (8) | 6 (18) | 3 (14) | 2 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No